CLINICAL TRIAL: NCT07183878
Title: A Prospective, Multicenter, Randomized Controlled Study Comparing Venetoclax-Enhanced BUCY With Standard BUCY Conditioning in High-Risk AML and MDS Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Venetoclax-Enhanced BUCY vs. Standard BUCY Conditioning in High-Risk AML and MDS Patients Undergoing Allo-HSCT (Ven-BUCY Study)
Acronym: Ven-BUCY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Ruijin Hospital North Shanghai Jiao Tong University School of Medicine (Unknown)
Responsible Party: Principal Investigator, Yanmin Zhao, Dr, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ven-BUCY
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; High-Risk Acute Myeloid Leukemia; Myelodysplastic Syndromes; High-Risk Myelodysplastic Syndromes
Keywords: Venetoclax; BUCY conditioning; Allogeneic Hematopoietic Stem Cell Transplantation; Myeloablative Conditioning; Relapse-Free Survival; Graft-versus-Leukemia; GVHD; High-Risk AML; High-Risk MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by disease (AML vs. MDS) and randomly assigned in a 1:1 ratio to receive either Venetoclax-enhanced BUCY conditioning or standard BUCY conditioning prior to allo-HSCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vene-BUCY (Experimental): Participants in this arm will receive a venetoclax-enhanced BUCY conditioning regimen before undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT). Venetoclax is administered from day -14 to -8 (400 mg/day for patients ≥14 years; 360 mg/m²/day for patients aged 12-14 years). Standard BUCY regimen includes busulfan (0.8 mg/kg every 6 hours, days -7 to -4), cyclophosphamide (60 mg/kg/day, days -3 and -2), and MeCCNU (250 mg/m² on day -1). Antithymocyte globulin (ATG) may be added for donor or recipient age >40 years. Venetoclax dose is reduced if co-administered with strong CYP3A4 inhibitors such as posaconazole.
  Interventions: Drug: Venetoclax
- BUCY (Active Comparator): Participants in this arm will receive the standard BUCY myeloablative conditioning regimen prior to allo-HSCT. The regimen includes busulfan (0.8 mg/kg every 6 hours, days -7 to -4), cyclophosphamide (60 mg/kg/day, days -3 and -2), and MeCCNU (250 mg/m² on day -1). ATG may be included in cases where the donor or recipient is over 40 years old. No venetoclax is used in this arm.
  Interventions: Other: None-placebo

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is administered orally at 400 mg/day for participants ≥14 years or 360 mg/m²/day for those aged 12-14 years, from day -14 to -8 before allogeneic hematopoietic stem cell transplantation (allo-HSCT). Dose is adjusted to 100 mg/day (or 90 mg/m²/day for pediatric patients) if used with strong CYP3A4 inhibitors such as posaconazole.
  Other Names: ABT-199; Venclexta
  Arms: Vene-BUCY
Other: None-placebo — Participants in this arm will not receive venetoclax as part of their conditioning regimen. They will undergo standard myeloablative conditioning with BUCY (busulfan, cyclophosphamide, and MeCCNU), prior to allogeneic hematopoietic stem cell transplantation. This arm serves as the active comparator to evaluate the addition of venetoclax in the experimental arm.
  Arms: BUCY

SUMMARY:
This is a prospective, multicenter, randomized controlled trial designed to evaluate the efficacy and safety of venetoclax-enhanced BUCY (Ven-BUCY) conditioning compared to the standard BUCY regimen in patients with high-risk acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS) undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT). Eligible participants aged 12 to 60 years will be randomized 1:1 to receive either Ven-BUCY or standard BUCY conditioning. The primary endpoint is relapse-free survival (RFS) at two years post-transplant. Secondary outcomes include overall survival, relapse rate, non-relapse mortality, measurable residual disease (MRD), and treatment-related adverse events. The study aims to improve post-transplant outcomes by deepening disease remission through the addition of venetoclax, a BCL-2 inhibitor known to target leukemia stem cells and enhance chemotherapy sensitivity.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains the only curative therapy for high-risk acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS). However, post-transplant relapse remains the leading cause of treatment failure, especially among patients receiving matched sibling or unrelated donor transplants. While myeloablative conditioning (MAC) regimens like BUCY (busulfan + cyclophosphamide) offer stronger anti-leukemic effects compared to reduced-intensity regimens, the relapse rate in high-risk myeloid neoplasms remains unacceptably high, partly due to residual leukemia stem cells (LSCs).

Venetoclax, a selective BCL-2 inhibitor, has shown synergistic effects when combined with hypomethylating agents or intensive chemotherapy. It improves remission depth and targets chemotherapy-resistant LSCs. Emerging data suggest that venetoclax may also enhance graft-versus-leukemia (GVL) effects without significantly increasing the risk of graft-versus-host disease (GVHD).

This investigator-initiated, open-label, two-arm, randomized controlled trial will enroll 138 patients aged 12-60 years with high-risk AML or MDS across six transplant centers in China. Patients will be stratified by disease (AML vs. MDS) and randomized (1:1) to receive either:

Standard BUCY regimen: Busulfan (0.8 mg/kg q6h on day -7 to -4), Cyclophosphamide (60 mg/kg/day on day -3 and -2), and MeCCNU (250 mg/m² on day -1), with optional ATG for donors/recipients >40 years.

Ven-BUCY regimen: Venetoclax (400 mg/day or 360 mg/m²/day from day -14 to -8) in addition to the standard BUCY components, with similar ATG guidance. Antifungal prophylaxis and venetoclax dose adjustment (e.g., to 100 mg with posaconazole) will follow local guidelines.

Patients will be followed weekly during the first month post-transplant, monthly for 6 months, and every 3 months thereafter until 3 years post-enrollment. The primary endpoint is 2-year relapse-free survival (RFS). Secondary endpoints include overall survival (OS), non-relapse mortality (NRM), relapse rate, MRD clearance, and adverse events graded by CTCAE v5.0.

This study seeks to determine whether adding venetoclax to a standard myeloablative regimen can enhance anti-leukemic efficacy and improve long-term outcomes without increasing transplant-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) according to 2022 WHO classification
* Age between 12 and 60 years
* High-risk MDS as defined by at least one of the following:

  * IPSS intermediate-2/high risk or IPSS-R intermediate/high/very high risk
  * TP53 mutation
  * RAS pathway mutation (e.g., NRAS, KRAS, PTPN11, CBL, NF1, RIT1, FLT3, KIT)
  * Therapy-related MDS
* High-risk AML as defined by at least one of the following:

  * TP53, RUNX1, or ASXL1 mutation
  * t(6;9)(p23;q34.1)/DEK-NUP214
  * KMT2A rearrangement
  * BCR-ABL1 fusion
  * inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2)
  * -5/del(5q), -7, -17/abn(17p)
  * Complex or monosomal karyotype
  * FLT3-ITD high with wild-type NPM1
  * Initial WBC ≥ 10×10^9/L
  * Secondary AML with history of MDS/MPN or therapy-related AML
  * AML with specific mutations (SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, EZH2, BCOR, STAG2)
  * MRD positive before transplantation
* For AML: must have achieved CR or CRi prior to transplantation; for MDS: bone marrow blasts < 20%
* Availability of a matched related or unrelated donor (10/10 or 9/10 HLA match)
* ECOG performance status 0-2
* Creatinine clearance ≥ 60 mL/min (Cockcroft-Gault)
* AST/ALT ≤ 3 × ULN and total bilirubin ≤ 2 × ULN
* LVEF ≥ 50% by echocardiogram
* Life expectancy > 8 weeks
* Willingness to use effective contraception methods during and for a specified period after the study
* Signed informed consent

Exclusion Criteria:

* Uncontrolled cardiovascular disease or New York Heart Association class III/IV heart failure
* Other severe comorbid conditions that may interfere with study participation
* Known HIV infection or uncontrolled active hepatitis B or C
* Pregnant or breastfeeding women
* More than one prior hematopoietic stem cell transplantation
* Inability to understand the study protocol or provide informed consent
* History of grade ≥ 3 non-hematologic adverse reaction to prior venetoclax therapy
* Receipt of chemotherapy (except hydroxyurea/dexamethasone) or radiotherapy within 14 days before study treatment
* Ongoing use of BCR-ABL1, IDH, or FLT3 inhibitors without proper washout (≥ 7 days)

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2028-08-20 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) | From the date of transplantation until relapse or death from any cause, assessed up to 24 months
  Relapse-Free Survival (RFS) is defined as the time from the date of allogeneic hematopoietic stem cell transplantation (allo-HSCT) to the first documented relapse of the primary disease or death from any cause, whichever occurs first. Participants who remain alive and relapse-free will be censored at the time of last follow-up.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 36 months post-transplantation
  Overall survival (OS) is defined as the time from the date of transplantation to death from any cause. Patients who are alive at the last follow-up will be censored. Survival curves will be estimated using the Kaplan-Meier method.
Non-Relapse Mortality (NRM) | Up to 36 months post-transplantation
  Non-relapse mortality (NRM) is defined as death from any cause other than disease relapse after transplantation. Competing risk analysis will be used to assess NRM incidence between groups.
Relapse Rate | Up to 36 months post-transplantation
  Relapse rate refers to the cumulative incidence of disease recurrence post-transplantation, assessed through bone marrow evaluation, flow cytometry, and molecular markers. Competing risk models will be applied for statistical analysis.
Measurable Residual Disease (MRD) Status | Assessed monthly during the first 6 months, and then every 3 months until 24 months post-transplantation
  MRD will be assessed by multiparameter flow cytometry and/or molecular techniques at scheduled timepoints after transplantation to evaluate minimal residual leukemia. MRD positivity and conversion dynamics will be compared between groups.
Treatment-Related Adverse Events | From start of conditioning until 28 days after transplantation, and during follow-up up to 3 months
  Incidence and severity of treatment-related adverse events, including hematologic and non-hematologic toxicities, will be evaluated and graded according to NCI-CTCAE v5.0. Events will be compared between the VEN-BUCY and BUCY groups.
Incidence of Acute Graft-versus-Host Disease (aGVHD) | From day of stem cell infusion to day 100 post-transplantation
  Acute GVHD will be assessed and graded based on MAGIC (Mount Sinai Acute GVHD International Consortium) criteria. The cumulative incidence of grade II-IV and grade III-IV aGVHD will be compared between the VEN-BUCY and BUCY groups.
Incidence of Chronic Graft-versus-Host Disease (cGVHD) | From day 100 post-transplantation to 36 months
  Chronic GVHD will be evaluated according to the 2014 NIH consensus criteria. The cumulative incidence of overall and moderate-to-severe cGVHD will be recorded and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yanmin Zhao, MD, Principal Investigator — Bone Marrow Transplantation Center, The First Affiliated Hospital, Zhejiang University School Of Medicine
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol